CLINICAL TRIAL: NCT03566134
Title: A Therapeutic Exploratory Clinical Study to Evaluate the Efficacy and Safety of DA-8010 in Patients With Overactive Bladder
Brief Title: A Therapeutic Exploratory Clinical Study of DA-8010 in Patients With Overactive Bladder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA8010_OAB_II
Record Dates: First submitted 2018-06-12; First posted 2018-06-21 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2018-07

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — DA-8010; Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): DA-8010 placebo + Solifenacin succinate placebo
  Interventions: Drug: DA-8010 Placebo; Drug: Solifenacin succinate placebo
- DA-8010 2.5mg (Experimental): DA-8010 2.5mg + Solifenacin succinate placebo
  Interventions: Drug: DA-8010 2.5mg; Drug: Solifenacin succinate placebo
- DA-8010 5mg (Experimental): DA-8010 5mg + Solifenacin succinate placebo
  Interventions: Drug: DA-8010 5mg; Drug: Solifenacin succinate placebo
- Solifenacin 5mg (Active Comparator): DA-8010 placebo + Solifenacin succinate 5mg
  Interventions: Drug: DA-8010 Placebo; Drug: Solifenacin 5mg

INTERVENTIONS:
Drug: DA-8010 Placebo — Participants receive placebo to match DA-8010 orally once a day.
  Arms: Placebo; Solifenacin 5mg
Drug: DA-8010 2.5mg — Participants receive DA-8010 2.5mg orally once a day.
  Arms: DA-8010 2.5mg
Drug: DA-8010 5mg — Participants receive DA-8010 5mg orally once a day.
  Arms: DA-8010 5mg
Drug: Solifenacin 5mg — Participants receive solifenacin 5 mg orally once a day.
  Arms: Solifenacin 5mg
Drug: Solifenacin succinate placebo — Participants receive placebo to match solifenacin 5 mg orally once a day.
  Arms: DA-8010 2.5mg; DA-8010 5mg; Placebo

SUMMARY:
A Therapeutic Exploratory Clinical Study to evaluate the efficacy and safety of DA-8010 in Patients with Overactive Bladder and to determine the optimal dose of DA-8010

ELIGIBILITY:
Inclusion Criteria:

Main Inclusion at Screening (Visit 1):

* Men and women 19 years or older with OAB symptoms for ≥ 3 months.
* Subject who is willing and able to complete the micturition diary correctly.
* Subject who is willing and able to provide informed consent indicating that they understand the purpose and procedures required for the study

Exclusion Criteria:

* Clinically significant Stress urinary incontinence or Mixed urinary incontinence where stress is the predominant factor
* Diagnosed with interstitial cystitis or bladder pain syndrome
* Clinically significant pelvic organ prolapse
* Subject who has neurologic status which is able to effect vesical function, such as multiple sclerosis, Spinal Injury or Parkinson's disease
* Medical history of malignant tumor in urinary system or pelvic organs
* Clinically significant bladder outlet obstruction or more than 200mL of post-void residual volume

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2019-12-27 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in mean number of micturitions per 24 hours | 12 weeks
  Change from baseline to Week 12 in mean number of micturitions per 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided